CLINICAL TRIAL: NCT03176576
Title: Patient Navigation in the Adolescent and Young Adult (AYA) Cancer Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-18420
Record Dates: First submitted 2017-06-02; First posted 2017-06-05 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Cancer
Keywords: cancer among adolescents; cancer among young adults; adolescents and young adults (AYA); quality of life; reduce stress; patient navigation; questionnaire; supportive care; distress levels; support resources; satisfaction survey; teen cancer
MeSH Terms: conditions — Neoplasms | interventions — Patient Navigation; Dental Assistants; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigator (PN) (Experimental): Patient Navigator (PN) Intervention Group. In addition to the Baseline Questionnaire and the Follow-up Questionnaire, PN intervention participants will complete a brief Patient Navigator Satisfaction Survey.
  Interventions: Behavioral: Patient Navigator (PN); Other: Baseline Questionnaire; Other: Follow-up Questionnaire; Other: Patient Navigator Satisfaction Survey
- Usual Care (UC) (Other): Usual Care (UC) Control Group. Control sample of patients not receiving PN intervention will complete a Baseline Questionnaire and the six-week Follow-up Questionnaire. Participants under UC will have access to all services typically provided to Moffitt Cancer Center (MCC) patients. Any baseline distress score greater than three will be reported to the patient's primary oncologist and clinic nurse.
  Interventions: Other: Baseline Questionnaire; Other: Follow-up Questionnaire

INTERVENTIONS:
Behavioral: Patient Navigator (PN) — Patient navigation (PN) is an intervention model designed to assist vulnerable patients in overcoming health system, personal and/or logistical barriers to care throughout the cancer care continuum. The strategic aims of PN are to reduce barriers and improve disease outcomes while also reducing distress and enhancing quality of life for the patient and family. Participants in the PN group will meet with a patient navigator.
  Other Names: assistant
  Arms: Patient Navigator (PN)
Other: Baseline Questionnaire — Complete a baseline questionnaire online or by meeting with a member of the study team. This questionnaire has items asking about the participant's health, distress levels, satisfaction with their care at Moffitt Cancer Center, and what support services they have used since their diagnosis. This questionnaire will take about 15 to 20 minutes of their time.
  Other Names: survey
Other: Follow-up Questionnaire — After participants complete the baseline questionnaire, they will be asked to complete a follow-up questionnaire approximately 6 weeks from when they completed the baseline questionnaire. The follow-up questionnaire will take about 15 to 20 minutes to complete.
  Other Names: survey
Other: Patient Navigator Satisfaction Survey — Evaluation of Patient Navigator intervention process.
  Other Names: satisfaction survey
  Arms: Patient Navigator (PN)

SUMMARY:
The purpose of this study is to develop and test a model of patient navigation that investigators hope will address the unique needs of adolescent and young adult (AYA) cancer patients and their families by minimizing barriers in their care and potentially improving the outcomes of their treatment while reducing distress and enhancing quality of life. Investigators plan to achieve this by increasing access to, and use of, the resources available at Moffitt Cancer Center for AYA patients and their families.

DETAILED DESCRIPTION:
Up to 80 participants may be recruited to this study at Moffitt Cancer Center to obtain a final sample size of 60 completed participants.

Participants will be identified in consultation with the patient's primary oncologist and program social worker. A research assistant (RA) will verify eligibility and consent eligible patients.

After completing a baseline questionnaire, participants will be randomly placed into one of two groups. Both groups will receive their normal care, but one group will also meet with a patient navigator. Participants in both groups will be asked to complete a follow-up questionnaire approximately 8 to 10 weeks from when they complete the baseline questionnaire. The follow-up questionnaire will take about 15 to 20 minutes to complete.

Participation in the study will last about 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 39 years old.
* Will undergo chemotherapy and/or radiotherapy and/or surgery with no plans to undergo a transplant procedure within the next 3 months.
* Have no previous cancer history other than non-melanoma skin cancer.
* Able to speak and read English.
* Able to provide written informed consent.

Exclusion Criteria:

* Does not meet any of the Inclusion Criteria.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Rate of Satisfaction with Patient Navigator | Upon completion of follow-up questionnaires and satisfaction surveys - up to 24 months
  Rate of participants reporting satisfaction with the patient navigator service, based on survey response scores.

SECONDARY OUTCOMES:
Rate of Improved Questionnaire Scores | Upon completion of follow-up questionnaires and satisfaction surveys - up to 24 months
  Follow-up Questionnaire scores for Patient Navigator group vs. Control group, as compared to Baseline Questionnaire Scores. Distress Indicator: Rating of 0 to 10, with 0 being No Distress and 10 being Extreme Distress). Health and Well Being Rating Categories: General health; Activity limitations; Problems with regular activities; Frequency of physical or emotional problems. Satisfaction with Care: Rating of 1 to 5, with 1 being Strongly Disagree and 5 being Strongly Disagree for 29 questions. Service Use: Regarding information and informational resources provided at Moffitt Cancer Center.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Donovan, PhD, MBA, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/